CLINICAL TRIAL: NCT03286595
Title: Smartphone Applications For Use in Youth With Early Psychosis in Community Outpatient Settings
Brief Title: Smartphone Applications Youth With Early Psychosis in Community Outpatient Settings
Acronym: BHCOEMobi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 782574
Record Dates: First submitted 2017-07-24; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Psychosis; Clinical High Risk for Psychosis
Keywords: early psychosis; clinical high risk; mobile health
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Psychosis (EP) (Experimental): EP participants will be individuals who are either a) at clinical high risk (CHR) for developing psychosis and/or bipolar disorder, or b) First Episode Psychosis (FEP) participants meeting criteria for schizophreniform disorder, schizophrenia, schizoaffective disorder or another psychotic, non-schizophrenia diagnosis including those with bipolar disorder.
  Interventions: Other: Mobi mHealth app
- Clinicians (Experimental): Clinicians/treatment team members who are providing treatment services to the EP participants at one of the three early psychosis clinics.
  Interventions: Other: Mobi mHealth app

INTERVENTIONS:
Other: Mobi mHealth app — Mobile application (i.e. the "app") that patients interact with via their smartphone to collect daily and weekly survey information. Data is visualized on a clinician-facing Dashboard, which can be used to inform treatment.

SUMMARY:
The project aims to test the utility of implementing a mobile health application ("mhealth app") in early psychosis care in the community outpatient setting and in the university medical center setting. We will enroll 60 individuals in the early stages of psychotic illness who are receiving care in two UC Davis affiliated community based early psychosis outpatient programs: the Aldea Child and Family Services SOAR Programs in Napa and Solano Counties (Napa SOAR, and Solano SOAR), as well as the UC Davis Early Psychosis Programs (EDAPT and SacEDAPT clinics). Early psychosis (EP) participants will include individuals at high risk for developing a psychotic illness (termed "clinical high risk" or CHR) and individuals within two years of their first psychotic episode (termed "first episode psychosis" or FEP). Over the course of five months, EP participants will use the app on their mobile device to complete daily surveys assessing mood, social interactions and medication adherence, and weekly surveys assessing clinical symptoms, sleep and medication adherence. EP participants will also complete clinical assessments with UC Davis research staff at the initial and final study appointments (baseline and five month timepoints). Clinicians working in the three early psychosis programs will also participate in the study. In their clinical role, they will interact with EP participants' app data via the Dashboard, a secure web-based portal, and provide feedback on the clinical utility of the data that is provided on the dashboard. EP participants and their clinicians will also provide feedback on the impact of the app on the therapeutic relationship.

DETAILED DESCRIPTION:
Although remission of psychotic symptoms following a patient's first episode of psychosis is achievable through pharmacological and psychosocial treatment, 50% of patients relapse within two years; 80% relapse within five. Relapse, defined as a recurrence of positive psychotic symptoms, is associated with cumulative increases in levels of psychotic symptoms following recovery, decreased social and community functioning, decreased quality of life, and increased hospitalizations. Given the negative impact on patients and their families, and the increasing cost of services as a function of relapse, development of effective relapse prevention strategies is imperative. Predictors of relapse amenable to treatment include: 1) clinical factors such as an exacerbation of clinical symptoms indicative of impending relapse; 2) treatment engagement factors such as medication adherence and therapeutic alliance; and 3) functioning factors such social impairments. Using mobile health technology in a community based outpatient clinic, we propose to specifically address these three types of relapse predictor variables.

The mobile health application tested in this study provides a user interface and a provider interface. The user interface is the mobile application (i.e. the "app") that patients interact with via their smartphone. This is designed to be simple and easily accessible. The app gathers "active" data, i.e. self-report surveys, which the user is alerted to via notifications on their device. Active data are analyzed and summarized for each patient on the "Dashboard", a provider-facing web portal for accessing concise and relevant information about a patient. The Dashboard provides up-to-date information regarding a patient's survey responses. Providers then use this information to better inform treatment decisions.

Specific aims and associated hypotheses are as follows:

Aim 1: Determine the feasibility and acceptability of the mhealth app in a community based outpatient early psychosis population. Hypothesis a: EPs will show high utilization of the mhealth app and low dropout, as well as high satisfaction and endorsement of continued use of the app. Hypothesis b: Clinicians will report high satisfaction and endorsement of continued use of the app.

Aim 2: Identify mhealth data related to key patient outcomes to inform calibration of patient status alerts. Hypothesis: Reductions in phone calls/text messages and/or increases in self-reported ratings of basic symptoms will predict psychotic symptom flares, increased clinic utilization, psychiatric ER visits and hospitalizations.

Aim 3: Evaluate the effect of the mhealth app on medication adherence, therapeutic alliance, and insight. Hypothesis a: After five months of app use, patients will report improved medication adherence, therapeutic alliance with their clinicians, and insight into their illness. Hypothesis b: After five months of use, clinicians will report improved therapeutic alliance with their patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for EP and CHR participants are: age 13-30 years, English fluency, and receiving clinical care at one of three UC Davis affiliated early psychosis clinics in the Northern California region: 1) UC Davis Early Psychosis Program (SacEDAPT & EDAPT clinics); 2) Aldea Solano SOAR Program; 3) Aldea Napa SOAR program.
* CHR participants will have no history of psychosis and will demonstrate attenuated psychotic symptoms consistent with the Structured Interview for Prodromal Syndromes (SIPS), or genetic risk (first-degree relative with psychosis) in conjunction with a substantial drop in functioning over the past year.
* FEP participants will be ascertained within three years or less from illness onset and have diagnoses of affective (i.e. bipolar) and non-affective psychosis (i.e. schizophrenia) according to DSM-IV criteria.

Exclusion Criteria:

* IQ below 70
* history neurological disorders
* current substance abuse/dependence

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility | 18 months
  Feasibility will be measured by utilization of the application (i.e. number of enrolled and active participants versus total patient population invited).
Acceptability/Satisfaction | 18 months
  Acceptability will be measured with satisfaction survey ratings of mhealth app by patients and clinicians.
Brief Psychiatric Rating Scale (BPRS) | 18 months
  a 24-item semi-structured clinical interview rating symptom severity at ascertainment across four domains: positive symptoms, negative symptoms, agitation/mania, and depression/anxiety.
Critical incidents | 18 months
  Includes information from patient chart: increased clinic contact, psychiatric ER visits or hospitalizations, and progression from a high risk state to first episode psychosis.
The Clinical Global Impression-Schizophrenia scale (Haro et al., 2003) | 18 months
  is a brief 12-item scale assessing illness severity and degree of improvement over follow-up that is appropriate for use in clinical or research settings.

SECONDARY OUTCOMES:
Medication adherence | 18 months
  The MARS (Thompson et al., 2000) is a 10-item self-report questionnaire assessing medication taking behavior, attitudes to medication, and side effects.
Therapeutic Alliance | 18 months
  Therapeutic alliance will be assessed with the STAR (Mcguire-Snieckus et al., 2007), a 12-item questionnaire with patient and clinician versions assessing positive collaboration and positive clinician input (both versions), non-supportive input (patient version), and emotional difficulties (clinician version).
Insight | 18 months
  Patient's insight into their illness will be assessed using the IS (Birchwood et al., 1994), an 8-item self-report questionnaire assessing awareness of illness, need for treatment, and attribution of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Imaging Research Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided